CLINICAL TRIAL: NCT01000129
Title: Adaptive - Predictive Planning for Hypofractionated Bladder Radiotherapy
Brief Title: Adaptive Planning in Bladder Cancer
Acronym: APPLY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Dr. Robert Huddart, Royal Marsden NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CCR3122
Record Dates: First submitted 2009-10-16; First posted 2009-10-22 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Bladder Cancer
Keywords: Radiotherapy; Bladder cancer; Adaptive planning
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Adaptive-Planning Organ Localisation (A-POLO) (Planning CT scan) — Planning CT scan performed by qualified planning radiographers
Other: Cone beam CT acquisition — Cone beam CT acquisition performed by therapy radiographers who have training and experience of using cone beam CT.

SUMMARY:
To demonstrate that radiotherapy treatments for bladder cancer can be delivered with greater accuracy using a new planning method and that this method can be used simply and effectively by those delivering treatment.

DETAILED DESCRIPTION:
This study integrates a novel adaptive planning methodology, Adaptive-Planning Organ LOcalisation (A-POLO), with optimised margins and cone beam CT technology for improving the accuracy of radiotherapy treatment delivery.

The previous study (CCR2873, REC 07/Q0801/13) evaluated the use of cone beam CT in radiotherapy for bladder cancer. A larger than expected number of bladder radiotherapy treatments were seen to have been delivered with some element of geographic miss. Using the novel adaptive planning method these fractions of radiotherapy could have been correctly treated. The feasibility of this method has been proven in the previous study, particularly it has been shown that this method is appropriate and provides a simple solution to the problem. It can be carried out by the radiographers at the treatment unit without adding extra time to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Histologically confirmed invasive carcinoma of the bladder
* Patient planned to receive hypofractionated radiotherapy to the bladder.
* No previous pelvic radiotherapy
* Written informed consent given according to ICH/GCP and national/local regulations.

Exclusion Criteria:

* Urinary catheter in situ: the presence of a urinary catheter degrades cone beam image quality and thus images would not be evaluable. Patients with a urinary catheter would not be expected to show variation in bladder filling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Assessment performed online at the treatment unit & verified offline by additional observer. Primary endpoint is met if there is greater than 75% concordance between the assessment made online & offline.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Robert Huddart, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom